CLINICAL TRIAL: NCT06702657
Title: A Randomized Clinical Trial on Urgent Angioplasty for IntraCranial Atherosclerotic Stenosis-related Large-Vessel Occlusion After Mechanical Thrombectomy (ICAS LVO-MT)
Brief Title: A Randomized Clinical Trial on Urgent Angioplasty for IntraCranial Atherosclerotic Stenosis-related Large-Vessel Occlusion After Mechanical Thrombectomy
Acronym: ICAS LVO-MT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Collaborators: The First People's Hospital of Changzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ICAS LVO-MT
Record Dates: First submitted 2024-11-21; First posted 2024-11-25 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: AIS; ICAS - Intracranial Atherosclerosis; Stroke
Keywords: ICAS; AIS; STROKE
MeSH Terms: conditions — Intracranial Arteriosclerosis; Stroke | interventions — Dosage Forms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Device: balloon dilatation and/or stenting
- Control group (Active Comparator)
  Interventions: Drug: medication

INTERVENTIONS:
Device: balloon dilatation and/or stenting — balloon dilatation and/or stenting immediately after randomization
  Arms: Intervention group
Drug: medication — medication after randomisation, mechanical thrombectomy again if necessary, avoiding balloon dilatation and/or stenting.
  Arms: Control group

SUMMARY:
A prospective, multicenter, randomized controlled, open-label, blinded outcome evaluation (PROBE) trial

DETAILED DESCRIPTION:
The main objective of AIS ICAS-MT study is to evaluate whether direct stenting, compared with medical therapy can benefit patients with acute ischemic stroke caused by CTA-confirmed large vessel occlusion (intracranial segments ICA, M1, BA, V4) who have been successfully recanalized by mechanical thrombectomy (MT) and are judged to be in situ ICAS lesions.

Primary outcomes: Functional recovery, defined as a sequence shift (improvement) in scores on the mRS at 90 (±14) days.

Secondary outcomes:

* Rate of good functional outcome (mRS of 0-2) at 90±14 days
* Rate of excellent functional outcome (mRS of 0-1) at 90±14 days
* Change in stroke severity (NIHSS score) at 24±12 hours
* Change in stroke severity (NIHSS score) at 7±2 days or discharge
* Proportion of target vessel recanalisation (eTICI≥2b) at 5±2 days confirmed by CTA
* Final infarct volume at 5±2 days
* EuroQol Five Dimensions (EQ-5D) Score at 90±14 days
* Barthel Index at 90±14 days
* mRS 3-6 at 90 days; Or stroke in the territory of the symptomatic intracranial artery (SIT) between 90 days and 365 days
* Stroke between 90 days and 365 days
* mRS Score shift at 365±30 days as an ordinal variable
* Rate of good functional outcome (mRS of 0-2) at 365±30 days
* Rate of excellent functional outcome (mRS of 0-1) at 365±30 days
* EuroQol Five Dimensions (EQ-5D) Score at 365±30 days
* Barthel Index at 365±30 days

Safety outcomes:

* Deaths within 90±14 days after enrolment
* Intracranial hemorrhage at 7 days post treatment or discharge (whichever occurs first)
* SAEs within 90±14 days after enrolment
* Any procedural complications
* The occurrence of new ischaemic stroke in the downstream territory of the occluded vessel within 90±14 days after enrolment
* Any cause of death within 365±30 days after enrolment
* Any occurrence of intracranial hemorrhage, subarachnoid hemorrhage, or intraventricular hemorrhage within 365±30 days after enrolment

ELIGIBILITY:
Inclusion Criteria:

Clinical inclusion criteria:

1. Age ≥ 18 years
2. National Institutes of Health Stroke Scale (NIHSS) score ≥6 before randomization
3. To receive mechanical thrombectomy <24 hours after AIS onset according to local guidelines
4. Signed informed consent form obtained from the subject (or approved surrogate)

Imaging inclusion criteria:

1. For subjects with anterior circulation stroke, ASPECTS ≥6 based on CT or DWI
2. For subjects with posterior circulation stroke, posterior circulation ASPECTS (pc-ASPECTS)≥6 and pons-midbrains index (PMI) < 3 based on CT or DWI

Angiography inclusion criteria:

1. The responsible occluded vessel is immediately recanalized (eTICI≥2b) after mechanical thrombectomy, ICAS is highly suspected and the focal residual stenosis of the main trunk is≥70%, and the responsible occluded vessels include the intracranial segment of the internal carotid artery, the M1 segment of the middle cerebral artery, the V4 segment of the vertebral artery, and the basilar artery
2. According to the judgment of the neurointerventional physician, the responsible artery is suitable for stenting angioplasty

Exclusion Criteria:

1. Pre-stroke mRS >2
2. Intracranial hemorrhage confirmed by CT before mechanical thrombectomy and enrolment
3. Suspected Intracranial hemorrhage after successful recanalization confirmed by 3D-CT
4. Tandem lesions: stenosis (or occlusion) of the extracranial segment of the internal carotid artery or vertebral artery combined with occlusion of large intracranial vessels, stenosis of intracranial arteries combined with occlusion of vessels distal to the stenosis
5. More than two severe stenosis of the responsible occluded vessel (internal carotid artery, middle cerebral artery, vertebral artery, and basilar artery)
6. Potential cardiac sources of emboli such as atrial fibrillation, left ventricular thrombus, heart valve replacement, atrial septal defect, ventricular septal defect, atrial myxoma, etc.
7. Current use of oral anticoagulants
8. Major surgery or serious trauma in the previous 2 weeks
9. Contraindication for mechanical thrombectomy or stenting angioplasty
10. Contraindication for antiplatelet treatment or allergy to contrast agent
11. History of gastrointestinal or urinary bleeding in the previous 3 weeks
12. Life expectancy less than 1 years
13. Current pregnant or breastfeeding status
14. Currently participating in another clinical trial that may affect the outcome assessment of this trial
15. Any other condition that, in the investigator's judgement, deems the individual unsuitable for enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 612 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2026-11-15 (Estimated); Study Completion 2027-08-15 (Estimated)

PRIMARY OUTCOMES:
Functional recovery | 90(±14) days
  defined as a sequence shift (improvement) in scores on the mRS

SECONDARY OUTCOMES:
Rate of good functional outcome | 90 (±14) days
  mRS of 0-2
Rate of excellent functional outcome | 90(±14) days
  mRS 0-1
Change in stroke severity (NIHSS score) | 24±12 hours
Change in stroke severity (NIHSS score) | 7±2 days or discharge
Proportion of target vessel recanalisation (eTICI≥2b) | 5±2 days
Final infarct volume | 5±2 days
EuroQol Five Dimensions (EQ-5D) Score | 90 (±14) days
Barthel Index | 90 (±14) days
mRS 3-6 at 90 days; Or stroke in the territory of the symptomatic intracranial artery (SIT) between 90 days and 365 days | 365days
  mRS 3-6 at 90 days; Or stroke in the territory of the symptomatic intracranial artery (SIT) between 90 days and 365 days
Stroke | between 90 days and 365 days
mRS Score shift | 365 (±30)days
Rate of good functional outcome | 365 (±30) days
  mRS of 0-2
Rate of excellent functional outcome | 365 (±30) days
  mRS of 0-1
EuroQol Five Dimensions (EQ-5D) Score | 365 (±30) days
Barthel Index | 365 (±30) days

OTHER OUTCOMES:
Deaths | within 90±14 days after enrolment
Intracranial hemorrhage | at 7 days post treatment or discharge (whichever occurs first)
SAEs | within 90±14 days after enrolment
Any procedural complications | Perioperative period
The occurrence of new ischaemic stroke in the downstream territory of the occluded vessel | within 90±14 days after enrolment
Any cause of death | within 365±30 days after enrolment
Any occurrence of intracranial hemorrhage, subarachnoid hemorrhage, or intraventricular hemorrhage | within 365±30 days after enrolment

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Liu, MD, PhD, Principal Investigator — Changhai Hospital

IPD SHARING:
Plan to Share IPD: Yes
Data can be shared with bona fide researchers after the publication of the main results, based on a submitted protocol to Oriental Collaboration group on Emerging Advanced therapy for Neurovascular diseases Consortium.
Supporting Information: Study Protocol, SAP
Time Frame: Data sharing will be available from 12 months after the publication of the main results.
Access Criteria: 1. The data sharing will be only for the purposes of health and medical research and within the constraints of the consent under which the data were originally gathered.
  2. The Custodian of the Collection will not consider any Proposals for data sharing that unblind, or potentially unblind, randomised comparisons in active / ongoing trials.
  3. Requesters should be employees of a recognised academic institution, health service organisation, commercial research organisation or from the pharmaceutical industry. Requesters must have experience in medical research.
  4. Requesters must be able to demonstrate through their peer review publications in the area of interest their ability to carry out the proposed use of the requested dataset from a Collection.
  5. The Requesters must not have a conflict of interest that may potentially influence their interpretation of any analyses.
URL: https://www.ocin.org.cn/